CLINICAL TRIAL: NCT02321631
Title: Efficacy of EPA-enriched Supplement Compared With Standard Formula on Body Weight Changing in Malnourished Head and Neck Cancer Patients Undergone Surgery: A Randomized Study
Brief Title: Efficacy of EPA-enriched Supplement in Malnourished Head and Neck Cancer Patients Undergone Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Kitti Jantharapattana, M.D., Assistant Professor, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC 57-073-13-1
Record Dates: First submitted 2014-12-04; First posted 2014-12-22 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Head and Neck Cancer
Keywords: Malnourished; Head and Neck Cancer; Surgery
MeSH Terms: conditions — Head and Neck Neoplasms; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EPA-enriched supplement (Experimental): EPA-enriched supplement is given to the patients for 3 weeks (1 week prior to surgery and 2 weeks post surgery). The supplement composes of 2.2 gm of EPA and 630 kcal daily.
  Interventions: Dietary Supplement: EPA-enriched supplement
- standard formula supplement (Placebo Comparator): The standard formula supplement is given to the patients for 3 weeks (1 week prior to surgery and 2 weeks post surgery). The supplement is 630 kcal daily without EPA.
  Interventions: Dietary Supplement: standard formula supplement

INTERVENTIONS:
Dietary Supplement: EPA-enriched supplement — EPA-enriched supplement is given to the patients for 3 weeks (1 week prior to surgery and 2 weeks post surgery). The supplement composes of 2.2 gm of EPA and 630 kcal daily.
  Arms: EPA-enriched supplement
Dietary Supplement: standard formula supplement — The standard formula supplement is given to the patients for 3 weeks (1 week prior to surgery and 2 weeks post surgery). The supplement is 630 kcal daily without EPA.
  Arms: standard formula supplement

SUMMARY:
The purpose of this study is to study the effects of EPA-enriched supplement compared with conventional supplement in malnourished head and neck cancer patients undergone surgery. Primary outcome is perioperative weight changing.

DETAILED DESCRIPTION:
To study the effects of EPA-enriched supplement compared with conventional supplement in malnourished head and neck cancer patients undergone surgery. The patients are divided into 2 groups receiving the different formula supplements. The both supplements are isocaloric. The patients receive the supplement for 3 weeks (1 week prior to surgery and 2 weeks post surgery) Primary outcome is perioperative weight changing. Secondary outcomes are body compositions, hospital stay days, complication and co-morbidity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as Head an Neck cancer with pathological confirmation
2. Receiving surgery as a primary treatment
3. Malnutrition screening tool(MST) is 2 or more

Exclusion Criteria:

1. Previously irradiated patient in the Head and Neck region
2. Previously receiving chemotherapy
3. Renal insufficiency with serum creatinine > 2.5 mg/dL
4. Liver function abnormality with total serum bilirubin > 3.0 mg/dL
5. Pregnancy

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-01; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Body weight at 3 weeks | 3 weeks
  Body weight measured in kilogram
Change from baseline in Body weight at 1 month | 1 month
  Body weight measured in kilogram
Change from baseline in Body weight at 3 months | 3 months
  Body weight measured in kilogram

SECONDARY OUTCOMES:
Change from baseline in fat-free mass percentage at 3 weeks | 3 weeks
  Percent of fat-free mass on the Bioelectrical Impedance Analysis (BIA)
Change from baseline in fat-free mass percentage at 1 month | 1 month
  Percent of fat-free mass on the Bioelectrical Impedance Analysis (BIA)
Change from baseline in fat-free mass percentage at 3 months | 3 months
  Percent of fat-free mass on the Bioelectrical Impedance Analysis (BIA)
Change from baseline in body fat percentage at 3 weeks | 3 weeks
  Percent of body fat on the Bioelectrical Impedance Analysis (BIA)
Change from baseline in body fat percentage at 1 month | 1 month
  Percent of body fat on the Bioelectrical Impedance Analysis (BIA)
Change from baseline in body fat percentage at 3 months | 3 months
  Percent of body fat on the Bioelectrical Impedance Analysis (BIA)

CONTACTS AND LOCATIONS:
Overall Officials: Kitti Jantharapattana, M.D., Principal Investigator — Faculty of Medicine, Prince of Songkla University
Locations (1):
- Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand